CLINICAL TRIAL: NCT07085169
Title: Low-dose Trifluridine/Tipiracil With Bevacizumab in Refractory Metastatic Colorectal Cancer: a Multicenter, Single-arm, Phase 2 Study
Brief Title: Low-dose Trifluridine/Tipiracil With Bevacizumab in mCRC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Jun Zhang, Clinical Professor, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAS-102/2025-No.412
Record Dates: First submitted 2025-07-16; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Colo-rectal Cancer; Third-line and Beyond Therapy; TAS 102; Bevacizumab
MeSH Terms: conditions — Colonic Neoplasms | interventions — Trifluridine; tipiracil; trifluridine tipiracil drug combination

STUDY DESIGN:
Intervention Model Description: All patients will receive low-dose trifluridine/tipiracil plus bevacizumab. Trifluridine/tipiracil will be given at a 17.5 mg/m2 dose orally twice daily in a 14-day cycle consisting of 10 treatment days/4 rest days. Bevacizumab will be given at a 5mg/kg dose intravenously once at day 1 in a 14-day cycle. This regimen will be administered until progression of disease, intolerable toxicity or withdraw of consent.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Trifluridine/tipiracil 17.5 mg/m2 bid. po. d1-10, q2w Bevacizumab 5mg/kg ivgtt. d1 q2w
  Interventions: Drug: Trifluridine/tipiracil (TAS-102) plus bevacizumab

INTERVENTIONS:
Drug: Trifluridine/tipiracil (TAS-102) plus bevacizumab — Trifluridine/tipiracil will be given at a 17.5 mg/m2 dose orally twice daily in a 14-day cycle consisting of 10 treatment days/4 rest days. Bevacizumab will be given at a 5mg/kg dose intravenously once at day 1 in a 14-day cycle. This is a single-arm study with all patients receiving these two drugs.

SUMMARY:
This is a phase II, single-center, prospective trial aimed to investigate the efficacy and safety of a modified regimen of trifluridine/tipiracil plus bevacizumab in refractory metastatic colorectal cancer. Patients will be treated with trifluridine/tipiracil (17.5 mg/m2 dose orally twice daily, d1-10, every 14-days) plus bevacizumab (5mg/kg dose intravenously once at day 1, every 14-days). The study treatment will be administered until progression of disease, intolerable toxicity or withdraw of consent.

DETAILED DESCRIPTION:
The treatment options as third-line therapy for metastatic colorectal cancer patients are limited. Trifluridine/tipiracil (TAS-102) plus bevacizumab has been approved in colorectal cancer for patients who are refractory to or intolerant of standard chemotherapy. However, the toxicity of trifluridine/tipiracil at standard dose a clinical concerned issue. Modifications of dose and treatment cycle of trifluridine/tipiracil have been investigated, and show promising effect to reduce the toxicity. In this study, patients with refractory metastatic colorectal cancer who have disease progression after at least 2 standard regimens will be treated with low-dose trifluridine/tipiracil plus bevacizumab. Trifluridine/tipiracil will be given at a 17.5 mg/m2 dose orally twice daily in a 14-day cycle consisting of 10 treatment days/4 rest days. Bevacizumab will be given at a 5mg/kg dose intravenously once at day 1 in a 14-day cycle. This regimen will be administered until progression of disease, intolerable toxicity or withdraw of consent.

ELIGIBILITY:
Inclusion Criteria:

1. age over 60 years old, male and female
2. histologically confirmed adenocarcinoma of the colon or rectum
3. patients with metastatic or advanced unresectable diseases who had received two or more previous chemotherapy regimens or intolerance to last regimen
4. with or without measurable lesions
5. ECOG 0 to 2, expected survival time over 3 months
6. Enough organ functions that can tolerate treatment: Absolute neutrophil count (ANC) ≥1.5x109/L, White blood count ≥3.5x109/L, Platelets ≥75x109/L, Hemoglobin (Hb) ≥80g/L, ALT/AST ≤2.5x ULN (for patient with liver metastasis ALT/AST ≤5x ULN), Serum bilirubin ≤1.5x ULN, Serum creatinine ≤1.5x ULN.
7. Signed informed consent and willing to follow the study protocol

Exclusion Criteria:

1. symptomatic metastases of central nervous system
2. other primary malignancies
3. uncontrollable comorbidities, such as hypertension, thrombotic diseases, chronic kidney disease
4. organ functions that cannot tolerate study treatment
5. bowel obstruction or other conditions affecting oral administration
6. allergic to study medication
7. other conditions that patients are unsuitable for this study assessed by the investigators

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
6-month progression-free survival rate | 6 months
  Defined as the proportion of patients who remain free from disease progression (as per RECIST criteria) or death for at least 6 months following initiation of study treatment.

SECONDARY OUTCOMES:
Adverse events | through study completion, an average of 1 year
Objective response rate | up to 16 weeks
Progression free survival | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
Overall survival | From date of enrollment until the date of death from any cause, assessed up to 100 months

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - SanMing First Hospital, Sanming
  - Ruijin Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided